CLINICAL TRIAL: NCT05713669
Title: Impact of Resident Participation in Post-ICU Follow Up Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jakob McSparron, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00225631
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Professional Burnout
Keywords: Perceptions of critical care; Professional fulfillment.
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: A Total of 20 residents will be recruited (10 residents in the intervention arm; 10 residents in the control arm). One resident in each pair will be randomized to participate in a follow up encounter in the post-ICU clinic with the patient that residents have cared for (intervention) and one will have no follow up encounter (control). There will be 10 patients enrolled for the study and will not be randomized into any arm. Outcomes are based on the residents only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Residents meet ICU patients during follow-up visit (encounter) (Experimental): Residents will be paired according to the patient that were cared.
  Interventions: Behavioral: Encounter visit with Patients
- Residents in the non-encounter group (Other): Residents will not meet with patients that were in the ICU.
  Interventions: Behavioral: Non-encounter surveys

INTERVENTIONS:
Behavioral: Encounter visit with Patients — Participants in this encounter group will be asked to complete a pre and post-intervention survey, participate in a meeting with a former ICU patient at a post-ICU clinic, and undergo an in-person interview within fourteen days following the encounter.
  Arms: Residents meet ICU patients during follow-up visit (encounter)
Behavioral: Non-encounter surveys — Surveys will be completed pre and post patient follow-up.
  Arms: Residents in the non-encounter group

SUMMARY:
This study is being conducted to describe the impact of a meeting between patients that were admitted to the intensive care unit (ICU) and a provider that cared for the patients during the period of critical illness. The study team is aiming to describe the effect this meeting has on the physician that previously cared for the patient.

The study team hypothesizes that facilitating involvement in post-ICU clinic and creating longitudinal relationships between providers of critical care and survivors of critical illness will have positive effects on trainees, both in professional fulfillment and burnout scores and in perceptions of critical care.

DETAILED DESCRIPTION:
Physicians and patients that had been cared for in the ICU will be enrolled in this project. Residents that are recruited will be randomized to the encounter group or the control group.

ELIGIBILITY:
Inclusion Criteria for Patients:

- Must be eligible for Post ICU Longitudinal Survivor Experience (PULSE) clinic follow up and/or have received referral to clinic

Inclusion criteria for Residents:

* Must have completed at least one 2-week rotation in the medical ICU at the University of Michigan
* Must have cared for an enrolled patient in the study

Exclusion Criteria for Patients:

- Died during ICU stay

Exclusion Criteria for Residents:

- Provided only "cross-cover" for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in the Professional Fulfillment Scale | Baseline (pre-post ICU follow-up visit), approximately 14 days post patient's follow-up visit
  The survey consists of 6 questions that are measured on a 5 point Likert scale (scored 0 to 4, with 4 representing higher fulfillment).
Changes in the Burnout Scale | Baseline (pre-post ICU follow-up visit), approximately 14 days post patient's follow-up visit
  This scale has 4 questions that will indicate the level of burnout with scores from not at all =0 - extremely =4. A higher score indicates a higher sense of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob McSparron, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No